CLINICAL TRIAL: NCT06997809
Title: ENDometriosis: Evaluation of Detection and Need for ALGOlogic Care Before Surgery
Acronym: ENDALGO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 87RI23_0049 (ENDALGO)
Record Dates: First submitted 2025-02-05; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis, Pain
Keywords: endometriosis, algologic care; pain, quality of life
MeSH Terms: conditions — Endometriosis; Pain | interventions — Critical Pathways

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Surgery without calculation of pain questionnaire scores
- group with adapted support (Experimental): The calculation of pain questionnaire scores is carried out to direct or not the patient towards pain consultations before surgery.
  Only patients with at least one positive test benefit from an algology consultation before surgery.
  Interventions: Other: pathway care

INTERVENTIONS:
Other: pathway care — Group for whom the test results will be used to determine the management strategy. If one of the tests performed before randomization is positive an algological consultation before surgery will be performed with an adapted treatment. Then surgical treatment as planned.
  If all tests are negative, surgical treatment is performed. The dedicated algology consultation must be done with an experienced practitioner different from the one who will perform the surgery. A rapid algological treatment circuit must be put in place to maintain the surgery date set.
  Group without using the results of test for associated pain components. Standard surgical treatment as planned through dedicated staff on endometriosis treatment.
  Arms: group with adapted support

SUMMARY:
Endometriosis surgery is required when medical treatment fails to release women from pain. However, complete surgery does not work every time to improve patients' symptoms. Algological care is one of the options to treat the pain before surgery and their related complications (neuropathy, sensitization, and catastrophism) that could be associated to nociceptive pain.

But not all patients could benefit from this pathway and no screening strategy does exist to detect these complications that could be treated prior to endometriosis surgery

ELIGIBILITY:
Inclusion criteria:

* Maternal age from 18 up to 50 years old (50 non included).
* Women affiliated to social coverage insurance
* Women who understand French
* Women who signed the written consent
* Women with impaired quality of life (pain) linked to endometriosis
* Women with formal radiological signs of endometriosis (MRI lesions more than 5 mm or endometrioma more than 20 mm on radiological examinations).
* Surgical indication for resection of lesions by laparoscopy or robotic surgery for management of pain or impairment of quality of life
* Patients requiring complete conservative or radical resections of all lesions
* Indication of surgery validated within dedicated meeting for endometriosis.
* Purpose of pain associated or not with infertility
* Date of surgery fixed with sufficient time for algological treatment. Maximum delay of 4 months between randomization and surgery

Exclusion criteria:

* Women undergoing surgery for the purpose of infertility
* Patient with previous surgery for removal of deep lesions of endometriosis or endometriotic cysts (history of exploratory laparoscopy accepted)
* Patient with suspicious lesions on MRI or specialized ultrasound.
* A patient who needs to be treated for another uterine pathology at the same time.
* Pregnant women
* Patient with a desire for pregnancy immediately and/or within one year after surgery
* Women who refuse clinical examination (some algological tests couldn't be performed without clinical examination)
* Patient who has already received algological treatment or who should receive it before surgery
* Patient with previous other psychiatric disorders (depressive symptoms treated)
* Women without rights

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life | 1 year after surgery
  Quality of life is assessed by the EHP5 score translated in French and validated in endometriosis. The primary endpoint is the comparison of EHP5 scores between the 2 groups (intervention vs. standard treatment) at 1 year after surgery for complete removal of deep endometriosis

SECONDARY OUTCOMES:
Evaluation of satisfaction | 6 months and 1 year after surgery
  Evaluation of satisfaction according to the CGI (Clinical Global Impression), at 6 months and 1 year
Evaluation of endometriosis-specific pain | From randomization to 6 months and 1 year
  Evaluation of endometriosis-specific pain according to the ENDOPAIN 4D score (which vary from 0 (no pain component) up to 110 (worst pain component)) before randomization and after surgery performed in all cases at 6 months and 1 year.
Evaluation of pain according to a Simple Numerical Scale (NSS) | 6 months and 1 year after surgery
  Evaluation of their score difference (2) and evaluation of pain according to a Simple Numerical Scale (NSS) ( from 0 (no pain) up to 10 (worst pain) before / after surgery at 6 months and 1 year
Improvement of EHP5 score | 6 months and 1 year after surgery
  Improvement of Endometriosis Health Profile (EHP5) score (from 0 (best quality of life) up to 100 (worst quality of life)) at 6 months and 1 year and difference between the beginning and between the two groups.
Assessment of prevalence of complex pain syndrome | Baseline
  Assessment of prevalence of complex pain syndrome in the whole population included: neuropathic pain (DN4 (from 0 (no symptoms) up to 10 (the most symptoms)) and PainDETECT score (from 0 (no probability of neuropathic pain unlikely) up to 38 (probability of neuropathic pain more likely)), sensitization (peripheral and central with Perineal Pain Sensitization Criteria (PPSC) (from 0 (no criteri) up to 10 (all criteria)) and Central Sensitization Inventory (CSI) score (from 0 ( no component) up to 100 (always and all components), associated catastrophizing (Pain Catastrophizing Score (PCS) (from 0 (no catastrophizing compenent) up to 52 (always and all catastrophizing components).
Assessment of determinant of complex pain syndrom of endometriosis | Baseline
  Assessment of determinants (previous medical conditions, demographical medical data and previous treatment before surgery) of complex pain syndrome of endometriosis (as describe in previous secondary outcome) with statistical modelization.
Calculation of the performance of the CSI test | Baseline
  Calculation of the performance (sensitivity, specificity, prevalence, accuracy) of the CSI test within this population.
Calculation of performance of each test and correlation | Baseline
  Calculation of the performance of each test proposed before randomization (DN4, PainDETECT, PPSC and PCS score) (prevalence) and correlation (kappa correlation) for neuropathic pain (DN4 and PainDETECT).

CONTACTS AND LOCATIONS:
Overall Officials: François Dr. Margueritte, Principal Investigator — University Hospital, Limoges
Locations (9):
- France (9):
  - Bordeaux University Hospital, Bordeaux, France
  - IFEMENDO, Bordeaux, France
  - Versailles Hospital, Le Chesnay, France
  - Saint-Vincent-de-Paul Hospital, Lille, France
  - Limoges University hospital, Limoges, France
  - Poissy-St-Germain Intercommunal hospital center, Poissy, France
  - Poitiers University Hospital, Poitiers, France
  - Mutual Clinic La Sagesse, Rennes, France
  - South Hospital Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided